CLINICAL TRIAL: NCT00704067
Title: Improving Work Outcomes for Veterans With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth W. Twamley, PhD, Principal Investigator, United States Department of Defense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT075291
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Traumatic Brain Injury
Keywords: vocational rehabilitation; supported employment; cognitive training; cognitive remediation; cognitive rehabilitation; veterans
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Employment, Supported; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Supported employment for 12 months plus cognitive training for the first 12 weeks
  Interventions: Behavioral: Supported employment plus cognitive training
- 2 (Active Comparator): Supported employment for 12 months plus one additional supported employment session per week for the first 12 weeks
  Interventions: Behavioral: Enhanced supported employment

INTERVENTIONS:
Behavioral: Supported employment plus cognitive training — Supported employment for 12 months plus cognitive training for the first 12 weeks
  Arms: 1
Behavioral: Enhanced supported employment — Supported employment for 12 months plus one additional supported employment session per week for the first 12 weeks.
  Arms: 2

SUMMARY:
The 12-month study will investigate a cognitive training augmentation of supported employment to improve cognitive performance and work outcomes, which are expected to result in improved quality of life and community integration for veterans with mild to moderate traumatic brain injuries. The primary hypothesis is that compared to veterans who receive enhanced supported employment, those who receive supported employment plus cognitive training will work more weeks during the 12 months.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF veteran
* History of mild-to-moderate TBI (loss of consciousness <6 hours; post-traumatic amnesia <7 days)
* Documented impairment in at least one neuropsychological domain
* Unemployed, but stating a goal of work
* Written informed consent to participate in the study

Exclusion Criteria:

* Current alcohol/substance abuse or dependence
* Participation in other intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Weeks worked | 12 months

SECONDARY OUTCOMES:
Hours worked | 12 months
Dollars earned from working | 12 months
Cognitive performance | 3, 6, and 12 months
Neurobehavioral symptoms | 3, 6, and 12 months
Quality of life | 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W Twamley, PhD, Principal Investigator — University of California, San Diego, VA San Diego Healthcare System, and Veterans Medical Research Foundation
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Derived] Walter KH, Jak AJ, Twamley EW. Psychiatric comorbidity effects on compensatory cognitive training outcomes for veterans with traumatic brain injuries. Rehabil Psychol. 2015 Aug;60(3):303-8. doi: 10.1037/rep0000049. Epub 2015 Jul 6. PMID 26147236